CLINICAL TRIAL: NCT00722670
Title: Woman-Focused HIV Prevention With Pregnant African-Americans
Brief Title: Pregnant Women's CoOp
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: RTI International (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Felicia A. Browne, ScD, MPH, Senior Research Social Epidemiologist, RTI International
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R01DA020852 (NIH); R01DA020852 (NIH)
Record Dates: First submitted 2008-07-23; First posted 2008-07-25 (Estimated); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: HIV
Keywords: risk reduction; prevention; HIV prevention
MeSH Terms: conditions — Risk Reduction Behavior | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Woman-focused (WF) (Experimental): Woman-focused intervention (Women's CoOp)
  Interventions: Behavioral: Woman-focused intervention
- Treatment as Usual (TAU) (Active Comparator): TAU (substance abuse treatment only)
  Interventions: Behavioral: Treatment as Usual

INTERVENTIONS:
Behavioral: Woman-focused intervention — Participants in this group received a four individual sessions of the woman-focused intervention, in addition to services that were part of their substance abuse treatment program
  Arms: Woman-focused (WF)
Behavioral: Treatment as Usual — Participants in this group only received services that were part of their substance abuse treatment program
  Arms: Treatment as Usual (TAU)

SUMMARY:
We will iteratively adapt and modify the NC woman-focused intervention (Women's CoOp), including the field manual and instrumentation, to focus on pregnant African-American women who abuse crack, are currently in substance abuse treatment, and are at risk for HIV or are HIV positive. We then will test the newly developed intervention in a Stage IB pilot-sized randomized clinical trial (RCT) in a traditional substance abuse treatment clinic to determine (a) feasibility; (b) relative efficacy compared with substance abuse treatment-as-usual (TAU), across several domains of functioning (e.g., substance use, HIV risk behaviors); and (c) the intervention's potential mechanisms of action.

The specific aims of this Stage IA/B study are as follows:

Aim 1. To adapt the culturally specific, manualized woman-focused intervention to specifically address issues of pregnancy and substance abuse, relationships with men, social support, parenting, HIV status, living with HIV, antiretroviral (ARV) treatment, and HIV risk-reduction methods for pregnant and postpartum women.

Aim 2. To compare the relative efficacy of the woman-focused intervention for pregnant women relative to standard substance abuse treatment to sustain reductions in substance abuse and sexual risk behaviors, maintain retention in drug treatment, reduce violence, and improve prenatal care and ARV treatment adherence (as needed) at 3- and 6-month follow-up.

Aim 3. To explore the intervention's potential mechanisms of action (e.g., by examining the mediating effects of changes in knowledge about HIV risk behaviors, psychological distress, readiness for change) and moderating factors (e.g., HIV status, age, stage of pregnancy, relationships with men) that may influence response to the treatment.

DETAILED DESCRIPTION:
We iteratively adapted and modified the NC woman-focused intervention (Women's CoOp), including the field manual and instrumentation, to focus on pregnant African-American women who abused crack, were currently in substance abuse treatment, and were at risk for HIV or were HIV positive. We then tested the newly developed intervention in a Stage IB pilot-sized randomized clinical trial (RCT) in a traditional substance abuse treatment clinic to determine (a) feasibility; (b) relative efficacy compared with substance abuse treatment-as-usual (TAU), across several domains of functioning (e.g., substance use, HIV risk behaviors); and (c) the intervention's potential mechanisms of action.

The specific aims of this Stage IA/B study were as follows:

Aim 1. To adapt the culturally specific, manualized woman-focused intervention to specifically address issues of pregnancy and substance abuse, relationships with men, social support, parenting, HIV status, living with HIV, antiretroviral (ARV) treatment, and HIV risk-reduction methods for pregnant and postpartum women.

Aim 2. To compare the relative efficacy of the woman-focused intervention for pregnant women relative to standard substance abuse treatment to sustain reductions in substance abuse and sexual risk behaviors, maintain retention in drug treatment, reduce violence, and improve prenatal care and ARV treatment adherence (as needed) at 3- and 6-month follow-up.

3. Estimated Enrollment: Can this be changed to 59 (the final enrollment)? Also, is there a way to change "Estimated" to "Final" or something more definite? 4. Study Start Date: Can this be changed to May 2007? 5. Study Completion: February 2009 (I know this date differs from the date in the email I sent earlier when I responded to your questions. Sorry, but this is the correct date to use) 6. Detailed Description: Can the current text be replaced with the following?

APPROACH: During Stage 1A, the team conducted a series of separate focus groups with an expert panel (including researchers, clinicians, and service providers); our Community Advisory Board; HIV+, substance-using, postpartum women; and HIV-, substance-using, postpartum women. We first inquired about how we could adapt the existing measures in the instrumentation, adapt the intervention to address issues of substance-using women who were pregnant, and determine the fidelity of its delivery. After this first set of focus groups, the Woman-Focused manual, measures, and intervention were revised to reflect new adaptations. Then the second set of focus groups with the same members were conducted for review of these materials and fidelity measures. Feedback was solicited to verify our adaptations and then it was pretested to further refine and finalize the manual and measures.

During Stage 1B, we recruited 59 women from treatment facilities in North Carolina. We marketed the study through a brochure as women entered the treatment programs. We also utilized existing outreach efforts for substance abusers at risk for HIV. Women who were eligible and consented to participate in the study gave a urine sample to assess drug use and take part in a 1½ hour ACASI interview. Topics included demographics, drug use, substance abuse treatment, physical health, sexual behavior, mental health, employment history, and criminal history. Once they completed the interview, the women were randomly assigned to either the women's intervention condition or a treatment as usual condition. Once randomized, women in the woman-focused intervention were asked to complete four one-hour intervention sessions within a month that included a personalized assessment and a personal action plan. As part of the second session, woman-focused intervention participants were offered HIV testing. Women in the TAU condition received the traditional substance abuse treatment services. Women in both groups were also assessed at 3-month and 6-month follow-up. Measures included behavioral outcomes, satisfaction with the intervention, and services received.

ELIGIBILITY:
Inclusion Criteria:

* Female
* 18 years of age or older
* Self-identify as Black/African-American
* Between 14 weeks (3½ months) and 32 weeks (8 months) gestation (pregnancy was confirmed via biological test)
* Self-report the use of an illicit drug within the past 12 months
* Currently enrolled in a substance abuse treatment program for at least 7 days
* Willing to provide written informed consent and verifiable locator information for follow-up assessments

Exclusion Criteria:

• Been in any previous CoOp studies

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2007-06; Primary Completion 2009-02 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
To compare the relative efficacy of the woman-focused intervention in reductions in substance abuse and sexual risk behaviors, maintain retention in drug treatment, reduce violence, and improve prenatal care and ARV treatment adherence (as needed). | 3- and 6-month follow-up

SECONDARY OUTCOMES:
To explore the intervention's potential mechanisms of action and moderating factors that may influence response to the treatment. | at 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Felicia Browne, ScD, Principal Investigator — RTI International
Locations (1):
- RTI International, Research Triangle Park, North Carolina, United States

REFERENCES:
- [Background] Wechsberg WM, Browne FA, Ellerson RM, Zule WA. Adapting the evidence-based Women's CoOp intervention to prevent human immunodeficiency virus infection in North Carolina and international settings. N C Med J. 2010 Sep-Oct;71(5):477-81. No abstract available. PMID 21473554
- [Background] Wechsberg WM, Browne FA, Poulton W, Ellerson RM, Simons-Rudolph A, Haller D. Adapting an evidence-based HIV prevention intervention for pregnant African-American women in substance abuse treatment. Subst Abuse Rehabil. 2011 Feb 10;2:35-42. doi: 10.2147/SAR.S16370. eCollection 2011. PMID 24474853
- [Background] Jones HE, Berkman ND, Kline TL, Ellerson RM, Browne FA, Poulton W, Wechsberg WM. Initial feasibility of a woman-focused intervention for pregnant african-american women. Int J Pediatr. 2011;2011:389285. doi: 10.1155/2011/389285. Epub 2011 Mar 23. PMID 21541069